CLINICAL TRIAL: NCT04211051
Title: Safety and Feasibility of a Novel Pulmonary Surgery Marker System in the Intraoperative Localization of Small Pulmonary Nodules
Brief Title: Safety and Feasibility of Pulmonary Surgery Marker System in the Intraoperative Localization of Small Pulmonary Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Futuo Zhida Medical Technology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Chair of thoracic department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTS-009
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Lung Neoplasms
Keywords: lung neoplasm; localization of lung nodules; ground glass opacity
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): LungBrella marker implanted into a predetermined position in the lung assisted by JediVision software and successfully marked the pulmonary nodules which needs to undergo Video-assisted thoracoscopic surgery
  Interventions: Device: LungBrella marker implantation and VATS partial lobe resection

INTERVENTIONS:
Device: LungBrella marker implantation and VATS partial lobe resection — The enrolled patients will receive a plain chest CT scan,then the data be loaded into JediVision software. The JediVision software can navigate the location of nodule and facilitate the implantation of LungBrella marker in the operating room after general anesthesia,then the patients will receive VATS partial lobe resection .

SUMMARY:
As the detection of small pulmonary nodules continuously grows, the intraoperative localization of small pulmonary nodules is in great demand. The intraoperative localization nowadays is usually done under local anesthesia before surgery. There is a certain rate of failure and complication. The result of our early animal experiments show that the pulmonary surgery marker system can deliver the intraoperative localization safely and precisely under anesthesia, and the average distance between the localization and the simulated lesion is less than 5mm during surgery. Therefore, the safety and feasibility of the system require further evaluation in patients

DETAILED DESCRIPTION:
This is a prospective, single-center clinical trial initiated by the investigator. LungBrella marker can be accurately implanted into a predetermined position in the lung assisted by JediVision software and successfully marked the pulmonary nodules which needs to undergo Video-assisted thoracoscopic surgery. The study is expected to enroll 10 patients. Finally, the effectiveness and safety of the method will be evaluated. This method not only can complete pulmonary nodule localization in the operating room without occupying the resources of radiology department, but also can let patients receive pulmonary nodule location after anesthesia. Thereby the risks during transportation are avoided and the suffering of patients is reduced.

ELIGIBILITY:
Inclusion Criteria:

Subjects should meet all of the following criteria

* diagnosis of pulmonary nodule, single nodule operation to be performed and nodule to be located by the decision of chief surgeon.
* commit to follow the research procedures and cooperate with the implementation of the whole process research
* 1 / 3 of pulmonary nodules are located in the periphery of the lung
* signed informed consent with date

Exclusion Criteria:

* the target lesion is close to the hilar or large blood vessels
* subjects with FEV1 less than 1.2 in lung function
* subjects with cardiac function III and cardiac function IV (NYHA, New York)
* subjects with uncontrollable acute pleura infection
* patients with previous history of thoracic surgery (thoracotomy), plural infection, and plural thickening and adhesion on the affected side
* Other factors that investigators disagree enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Positioning success rate | Immediately after resection
  When the distance between the LungBrella marker and the Pulmonary nodule is less than 10mm, the marker position is successful. The success rate is the proportion of successful cases to all operation cases

SECONDARY OUTCOMES:
Procedure time | Duration of procedure
  Collect total procedure time for lung localization and surgical resection.
Complications | One month
  Procedure-related complications will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hecheng Li, MD&PHD, Principal Investigator — Ruijin hospitalRuijin Hospital, Shanghai Jiao Tong University School of Medicine; Hecheng Li, MD&PHD, Study Chair — Ruijin Hospital
Locations (1):
- RuijinhospitalRuijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li C, Ji A, Jian Z, Zheng Y, Feng X, Guo W, Lerut T, Lin J, Li H. Augmented reality navigation-guided intraoperative pulmonary nodule localization: a pilot study. Transl Lung Cancer Res. 2023 Aug 30;12(8):1728-1737. doi: 10.21037/tlcr-23-201. Epub 2023 Aug 4. PMID 37691871
- [Derived] Li C, Zheng Y, Yuan Y, Li H. Augmented reality navigation-guided pulmonary nodule localization in a canine model. Transl Lung Cancer Res. 2021 Nov;10(11):4152-4160. doi: 10.21037/tlcr-21-618. PMID 35004246